CLINICAL TRIAL: NCT01170117
Title: Olanzapine vs Placebo for Outpatients With Anorexia Nervosa
Brief Title: Olanzapine Versus Placebo for Outpatients With Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Weill Medical College of Cornell University (Other); University of Pittsburgh (Other); Johns Hopkins University (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Evelyn Attia, Clinical Psychaitrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #6142/7117R; R01MH085921 (NIH)
Record Dates: First submitted 2010-07-23; First posted 2010-07-27 (Estimated); Results first posted 2017-08-25 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Anorexia Nervosa
Keywords: Eating Disorders; Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Control group receiving placebo
  Interventions: Drug: Placebo
- Olanzapine (Experimental): Group receiving olanzapine
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Dosing of olanzapine will begin at 2.5 mg and will be titrated to a maximum dose of 10 mg. The target dose of 10 mg of olanzapine was selected because published data from studies that used this dose indicated that it was helpful to patients.
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: Placebo — Control Group will receive placebo pill
  Arms: Placebo

SUMMARY:
Anorexia Nervosa (AN) is a serious illness associated with substantial morbidity and mortality. Weight restoration is a treatment priority, and better treatments are needed.

DETAILED DESCRIPTION:
This study is a 16-week randomized, double-blind, placebo-controlled trial of olanzapine in adult outpatients with AN. 160 individuals with AN, ages > 18, will be randomly assigned to receive olanzapine or placebo for 16 weeks together with a medication management treatment. Primary outcomes will include weight gain as well as psychological symptoms known to be associated with AN, including obsessionality, mood, and anxiety.

This project is based on evidence from a recently completed 8-week pilot study comparing the efficacy of olanzapine to placebo in outpatients with AN (PI: Evelyn Attia, MD), as well as a recently published 12-week trial of olanzapine vs placebo (Bissada et al, Am J Psychiatry, 2007) in which outpatient treatment with olanzapine was associated with weight improvement, improved psychological status, and no untoward metabolic effects among low-weight patients.

The investigators hypothesize that among underweight adult outpatients with AN receiving olanzapine vs. placebo, together with medication management treatment: 1)patients with AN receiving olanzapine will gain weight at a faster rate than those receiving placebo; and 2) patients with AN receiving olanzapine will demonstrate greater reduction in psychological symptoms, including obsessionality, mood, anxiety and eating disorder symptoms, than those receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Anorexia Nervosa
* Body Mass Index (BMI) between 14.0 and 18.5 kg/m2
* Between 18-75 years old
* Patient not pursuing intensive treatment (inpatient or day treatment) for weight restoration if BMI less than 18 kg/m2
* serum potassium > 2.5 mEq/L

Exclusion Criteria:

* Any medical or psychiatric problem requiring medical or psychiatric attention, significant metabolic disturbance upon psychiatrist presentation, and/or significant co-morbid illnesses that are not likely to benefit from proposed treatments or that need specialized treatments for non-eating disorder symptoms.
* Diabetes mellitus
* QTc > 480 msec at baseline or increase in QTc of > 35 msec since baseline ECG
* Significant hyperlipidemia (cholesterol, triglycerides > 1.5 x upper limit of normal)
* Current diagnosis of substance abuse or dependence
* Diagnosis of schizophrenia, schizophreniform disorder, bipolar illness (type I)
* Presence of movement disorder, tardive dyskinesia
* History of seizure disorder
* Dementia (subjects over age 55 will be assessed by an MMSE administered by a psychiatrist; those who receive an MMSE score >25 will be excluded)
* Allergy to olanzapine
* Documented treatment with 10 mg/day olanzapine x 8 weeks or known inability to tolerate olanzapine 10 mg/day
* Taking psychotropic (antidepressant, antianxiety, mood stabilizer, antipsychotic) medication within the 4 weeks prior to randomization, other than stable dose of Selective Serotonin Reuptake Inhibitor (SSRI) or Serotonin/Norepinephrine Reuptake Inhibitor (SNRI), or use of benzodiazepine or non-benzodiazepine sleep agents. These permissible medications may be continued during the trial if they have been in use by the patient for a period of > 4 weeks at an unchanged dose without any evidence of consistent weight gain (i.e., > 3 lbs/months)
* Taking other medication within the last four weeks prior to randomization, known to affect weight (e.g., steroids)
* Participation in a psychotherapeutic intervention associated with consistent weight gain (i.e. > 3 lbs/month). (Subjects may participate in the study if they are receiving stable outpatient psychotherapy for the 4 weeks prior to randomization as long as there have been no changes in therapy intensity and the psychotherapy has not been associated with weight gain > 3 lbs over the previous 4 weeks. Subjects may also participate if they recently received partial weight restoration treatment in an intensive inpatient or day program as long as they can document that they have not consistently gained weight in their current treatment setting for the 4 weeks prior to baseline screening.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Attia, MD, Principal Investigator — New York State Psychiatric Institute
Locations (5):
- United States (4):
  - Johns Hopkins, Baltimore, Maryland
  - New York State Psychiatric Institute, New York, New York
  - Weill Cornell Medical Center, White Plains, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Bissada H, Tasca GA, Barber AM, Bradwejn J. Olanzapine in the treatment of low body weight and obsessive thinking in women with anorexia nervosa: a randomized, double-blind, placebo-controlled trial. Am J Psychiatry. 2008 Oct;165(10):1281-8. doi: 10.1176/appi.ajp.2008.07121900. Epub 2008 Jun 16. PMID 18558642
- [Derived] Attia E, Steinglass JE, Walsh BT, Wang Y, Wu P, Schreyer C, Wildes J, Yilmaz Z, Guarda AS, Kaplan AS, Marcus MD. Olanzapine Versus Placebo in Adult Outpatients With Anorexia Nervosa: A Randomized Clinical Trial. Am J Psychiatry. 2019 Jun 1;176(6):449-456. doi: 10.1176/appi.ajp.2018.18101125. Epub 2019 Jan 18. PMID 30654643

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from December 2010 through June 2016 at each of the five study sites, which are medical clinics: Columbia University-New York State Psychiatric Institute, Weill Cornell Medical College, Centre For Addiction And Mental Health in Toronto, University Of Pittsburgh and Johns Hopkins University.
Pre-assignment Details: A total of 25 individuals across sites discontinued the trial prior to group assignment, and 17 were withdrawn by investigators before randomization. These individuals were excluded from the trial due to various reasons such desiring alternate care, and not being interested in medication.
Period: Overall Study
Arm/Group | Placebo | Olanzapine
Started | 77 | 75
Completed | 47 | 55
Not Completed | 30 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Olanzapine | Total
Number analyzed (Participants) | 77 | 75 | 152
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.0 (10.9) | 28.0 (10.8) | 29.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 71 | 146
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 71 | 67 | 138
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 71 | 69 | 140
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 16.69 (1.18) | 16.79 (1.17) | 16.7 (1.20)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Weight Change
Description: Comparison of rate of weight change between patients receiving olanzapine and those receiving placebo
Time Frame: Weekly during 16-week trial and twice during 8 weeks follow-up
Population: Patients assigned to receive placebo or olanzapine for 16 weeks.
Measure: Mean (Standard Error); unit: kg/m^2 per month
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 77 | 75
kg/m^2 per month | 0.095 (0.053) | 0.260 (0.051)

2. Primary Outcome: Psychological Change
Description: Comparison of psychological change as measured by the Yale-Brown Obsessive Compulsive Scale (YBOCS), in patients receiving olanzapine compared with those receiving placebo. The Y-BOCS is divided into two sections: obsessive and compulsive. The scores for each section range from 1 to 20. The overall scores are obtained from adding scores for the two sections, to obtain a range between 2-40. A lower score reflects improvement/ fewer obsessive compulsive symptoms. A score of 25 or more is considered moderately severe, a score of 30 or more is considered severe, and a score of more than 35 is considered very severe.
Time Frame: Weekly during 16-week intervention and twice during 8-week follow-up
Measure: Mean (Standard Deviation); unit: YBOCs score units per month
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 77 | 75
YBOCs score units per month | 0.762 (0.375) | 0.800 (0.350)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 24 weeks of study participation (16 weeks of active participation, and 8 weeks of followup).
Arm/Group | Placebo | Olanzapine
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/75
Serious Adverse Events (participants affected / at risk) | 13/77 | 16/75
Other Adverse Events (participants affected / at risk) | 0/77 | 2/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=77) | Olanzapine (N=75)
Patient hospitalized in eating disorder center to pursue higher level of care. (Psychiatric disorders) | 7 (7) | 11 (11)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) — Patient exceeded the prescribed dose of olanzapine vs. placebo in anticipation of her week 8 olanzapine blood level laboratory test
Abnormal EKG (Cardiac disorders) | 1 (1) | 1 (1)
Physical injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) — Bone broken
Malignant mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Body spasm (Psychiatric disorders) | 1 (1) | 0 (0) — Patient admitted to the ER after experiencing "total body spasms" and was treated with fluids, Valium, and Benadryl. After an evaluation, study MD concluded that the participant may have had a dystonic reaction.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=77) | Olanzapine (N=75)
Mild undulating movement in his posterior tongue on the Abnormal Involuntary Movement Scale (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No